CLINICAL TRIAL: NCT03486444
Title: Exploring New and Next Generation Ultrasound Technologies for Medical Education, Patient Care, and New Indications
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: University of Cincinnati (Other)
Collaborators: Ohio Third Frontier (Other)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Professor, University of Cincinnati
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RP0509/2017H0356
Record Dates: First submitted 2018-02-21; First posted 2018-04-03 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Portable Ultrasound
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Patient population (Experimental): When a patient receives an ultrasound examination as part of standard of care or within another clinical research trial, such an examination may serve for an intra-individual comparator examination between conventional and new, ultra-portable ultrasound imaging. Patients will be identified in the clinical setting when appropriate and will be appropriately approached for consent for a combination of ultrasound with the physical exam, for medical student education, IV access, and novel application. Patients will be enrolled and accounted for in the appropriate sub-population.
  Interventions: Diagnostic Test: Phillips Lumify Diagnostic Ultrasound System; Other: Surveys
- Healthy volunteer population (Experimental): The volunteer population will allow us to practice the use of this equipment and understand the limitations and applicability. The results will be the images acquired as well as surveys from the volunteers and those performing the scans, who will be enrolled in the staff population of this study.
  Interventions: Diagnostic Test: Phillips Lumify Diagnostic Ultrasound System; Other: Surveys
- Student and staff population (Experimental): To understand the impact of ultraportable ultrasound, survey tools will be used to understand the workflow and clinical care applications and integration of these devices. All staff and student members will be appropriately consented; however, we anticipate that this portion of the study will be minimal risk.
  Interventions: Other: Surveys

INTERVENTIONS:
Diagnostic Test: Phillips Lumify Diagnostic Ultrasound System — portable ultrasound device
  Arms: Healthy volunteer population; Patient population
Other: Surveys — surveys assessing perception of ultrasound

SUMMARY:
This is a Phase I study to assess feasibility. There will be no impact on clinical care based on this study. The ultrasound system is FDA approved and could be used for clinical care independent of this research study. When a subject receives an ultrasound examination as part of standard of care or within another clinical research trial, such an examination may serve for an intra-individual comparator examination between conventional and new, ultra-portable ultrasound imaging. Patients will be identified in the clinical setting when appropriate and will be appropriately approached for consent for a combination of ultrasound with the physical exam, for medical student education, IV access, and novel application. Patients will be enrolled and accounted for in the appropriate sub-population. Additionally, to understand the impact of ultraportable ultrasound, survey tools will be used to understand the workflow and clinical care applications and integration of these devices. All staff and student members will be appropriately consented; however, the investigators anticipate that this portion of the study will be minimal risk with online consent waivers. Finally, the volunteer population will allow us to practice the use of this equipment and understand the limitations and applicability. The results will be the images acquired as well as surveys from the volunteers and those performing the scans, who will be enrolled in the staff population of this study. No significant risk is identified for subjects in this study. The largest risk, although still minimal, is an incidental finding. For this study, subjects will have the choice if they would like to be informed of an incidental finding. Reporting of incidental findings will be conducted by designated study staff after appropriate consultation and examination of the images by the PI or designee. While there are no direct benefits for subjects in this study, the study hopes to improve the implementation of ultrasound into the clinical setting into the future. This Phase I study aims to examine the feasibility of implementation and the impact on the clinical setting. Additionally, this study hopes to examine the utility and usefulness of ultrasound in medical education and thereby hopes to improve the physical exam skills of clinicians for the future.

DETAILED DESCRIPTION:
Ultrasound is a non-invasive, effective imaging methodology that is being used for many applications. The clinical availability of an ultra-portable app-based ultrasound system is a technology leap that has the potential to completely change the way ultrasound is used.

The objectives of this study are:

1. Evaluate feasibility of use of a new app-based ultra-portable, ultrasound system in the clinical setting
2. Review image quality and consistency of quality
3. Examine the use of new app-based ultra-portable ultrasound as an extension of the physical exam and implementation into medical education
4. Determine potential clinical applications, opportunities, and limits
5. Perform intra-individual comparison to current clinical use ultrasound device
6. Exam the perception and integration of new, ultra-portable ultrasound systems
7. Determine the potential educational value to medical student experience

Experimental activities performed as a part of this research study are divided into three different categories based on participant population: Patient population: For these patients, the non-research activities will be their standard of care ultrasound examination or their ultrasound examination within another clinical research trial. For these participants, the experimental activities could involve four different scenarios: 1) Patient having a standard of care US and participates in the comparator assessment using the new or ultra-portable US technology, 2) Patient having a physical examination by a medical student, resident or physician, 3) Patient requiring vascular access, 4) Patient has a medical diagnosis and within this clinical trial the investigators will use and evaluate the new ultrasound technology regarding its potential of enabling novel application. For each of these scenarios, in addition to the investigational ultrasound examination, the patient will be given a questionnaire to give feedback from his or her perspective. Staff population: For the staff population, research activities will involve a questionnaire to provide feedback regarding the experience and perception of the ultraportable ultrasound technology at the completion of each ultrasound imaging session. Volunteer population: For these participants, all activities will be performed solely for the research study (i.e. there is no standard of care ultrasound examination). The investigators plan to have the volunteers involved in two different scenarios, which would all take place after informed consent has been given and documented: 1) Participation in a single ultrasound exam session, 2) Participation in multiple ultrasound exams and multiple operator sessions. In addition to receiving one or more ultrasound examinations, the volunteers will be asked to complete a questionnaire to provide feedback from his or her perspective regarding the ultraportable ultrasound technology.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects or patients greater than or equal to 18 years of age
* Patients who are capable of giving informed consent

Exclusion Criteria:

* Prisoners
* Participants incapable of giving informed consent, even if they have a power of healthcare attorney who is clearly identifiable and available for the consenting process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Image Quality | through study completion, an average of 1-3 years
  Assessing the benefit of portable ultrasound to improve the capabilities of ultrasound imaging
Perception of portable ultrasound | through study completion, an average of 1-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Knopp, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

DOCUMENTS (1):
  • Study Protocol (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT03486444/Prot_000.pdf